CLINICAL TRIAL: NCT04146623
Title: A Randomized Double-Blind, Placebo Controlled, Phase I Study of the Safety, Tolerability and Immunogenicity of a Live Attenuated H1N1 Vaccine in Healthy Individuals
Brief Title: Safety Study of Live Attenuated Influenza Vaccine, CodaVax, Delivered Via Intranasal Spray
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Codagenix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CODA01-002
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Influenza
Keywords: live-attenuated vaccine; influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Normal Saline Placebo (Placebo Comparator): Saline (0.9%)
  Interventions: Biological: Normal Saline Placebo
- CodaVax-H1N1 (Experimental): Live-attenuated influenza vaccine
  Interventions: Biological: CodaVax-H1N1 influenza vaccine

INTERVENTIONS:
Biological: CodaVax-H1N1 influenza vaccine — CodaVax-H1N1, a live attenuated vaccine (LAIV) strain based on the A/California/07/2009 (H1N1) influenza virus, administered once intranasally via a sprayer at a dose of 8 x10^5 plaque forming units (PFU).
  Arms: CodaVax-H1N1
Biological: Normal Saline Placebo — Saline (0.9%) administered intranasally via sprayer
  Arms: Normal Saline Placebo

SUMMARY:
This study is being conducted to assess the safety, tolerability, and immunogenicity of the live-attenuated CodaVax-H1N1 influenza vaccine as compared to normal saline placebo both administered via intranasal spray to healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Adult volunteers, aged 18 to 45 years (at the time of screening) in good general health in the opinion of the Medical Investigator or delegate, with no significant medical history and no clinically significant abnormal findings at screening.
2. Participants must use highly effective, double contraception from the Screening Visit and up to the Follow-up Visit (Day 30).
3. Must be willing to comply with the following conditions to prevent the spread of Genetically modified organisms (GMO) according the Office of Gene Technology Regulator (OGTR) Licence (DIR 144):

   1. Hygiene measures intended to prevent interpersonal transmission of study drug must be implemented, including but not limited to frequent handwashing with soap or hand disinfectant, respiratory hygiene and cough etiquette within 7 days following vaccination
   2. Blood, tissue or organs must not be donated within 7 days of vaccination
   3. Severely immunosuppressed persons who require a protective environment are not to be cared for by the participant within 7 days of vaccination
   4. Contact is not to be made with severely immunosuppressed persons who require a protective environment within 7 days of vaccination
   5. All tissues and materials used to collect respiratory secretions are to be sealed in a primary container and placed within a secondary container so that it is not accessible to children or animals for 7 days until it is returned to the study site for disposal, for 7 days within vaccination
4. Contact is not to be made with infants <6 months of age within 7 days of vaccination.
5. Adequate venous access in the left or right arms to allow collection of a number of blood samples.
6. Must be sero-susceptible ≤10 hemagglutination inhibition (HAI) titre to CA/07/2009 Influenza virus (pre-screen).
7. Laboratory Testing:

   1. Full blood examination and biochemistry within the laboratory defined normal range unless deemed not clinically significant by the investigator, however a small drop below the normal range for Absolute Neutrophil Count (ANC) may be acceptable as per investigator discretion;
   2. Urinalysis: Negative urine glucose, negative or trace urine protein, negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis within institutional range)
8. Able to communicate effectively with study personnel and considered reliable, willing and cooperative in terms of compliance with the protocol requirements
9. Participant does not intend to start or change an existing physical conditioning regimen prior to or during the study period
10. Participant has voluntarily given written informed consent to participate in the study (prior study entry)
11. Participant is available for the duration of the study

Exclusion Criteria:

1. Immunodeficiency (including HIV) or autoimmune disorder, or participant is currently taking drugs (excluding steroids, see exclusion criteria 16) or was undergoing a form of treatment within 3 months prior to study entry that affects the immune system, or participant is living with somebody with the same
2. Participant is not to have had Guillain-Barre Syndrome
3. Received blood or blood products in the 3 months prior to screening
4. Received another vaccine within 30 days before screening
5. Received another influenza vaccine from 2016 to present year
6. Participants with plans to travel to the Northern Hemisphere during the Screening period
7. Participated in another clinical study (involving any investigational product or device) within 60 days before screening
8. Suffered previous anaphylactic reaction to foods, vaccines, drugs or hymenoptera stings, or has a history of severe allergic reactions (e.g. clinically severe urticaria, asthma)
9. Participants with active asthma or a history of childhood asthma which was treated with corticosteroids.
10. Participants with a known egg allergy
11. If female, pregnant, planning to become pregnant, or lactating, or participants is living with somebody who is pregnant or lactating.
12. Participant has a history of, or current evidence at the time of screening of abuse of alcohol or any drug substance, licit or illicit, or current alcohol consumption is > 4 standard drinks (or equivalent) per day
13. History of any psychiatric illness or psychological disorder which may impair the ability to provide written informed consent or participate in the study
14. Current or history of significant neurological, cardiovascular, pulmonary (including asthma), hepatic, rheumatic, autoimmune, hematological, metabolic or renal disorder
15. Clinically significant abnormal laboratory value at screening as determined by the Investigator
16. Known or suspected impairment/alteration of immune function, including: Chronic use of oral steroids (equivalent to 20 mg/day prednisone ≥12 weeks /≥2 mg/kg body weight / day prednisone ≥2 weeks) within 60 days prior to Day 0 (use of inhaled, IN, or topical corticosteroids is allowed, unless used for the management of asthma - see exclusion criteria 9). Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥12 weeks /≥2 mg/kg body weight/day prednisone ≥ 2 weeks) within 60 days prior to Day 0. Or participant is living with somebody with the same
17. Unusual dietary habits and excessive or unusual vitamin intake likely, in the opinion of the Investigator, to affect safety parameters
18. Participant is sero-positive to hepatitis C virus or hepatitis B virus.
19. Body temperature (oral) ≥38.0ºC or acute illness within 5 days prior to vaccination
20. Any other significant finding that, in the opinion of the Investigator, would increase the risk of the individual having an adverse outcome from participating in this study
21. Participant is a member of the team or is related or in a dependent relationship with a member of the study team, as defined as the Sponsor or study site personnel

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-10-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Reactions to vaccine | 6 days
  Number of solicited local and systemic reactions for CodaVax-H1N1 and placebo
Adverse events (AEs) | 30 days
  Number of subjects with AEs for CodaVax-H1N1 and placebo
Serious adverse events (SAEs) | 180 days
  Number of subjects with SAEs for CodaVax-H1N1 and placebo

SECONDARY OUTCOMES:
HAI antibody titers against A/California/07/2009 | Day 0 and 30
  Geometric mean titers (GMT) of anti-A/California/07/2009 (H1N1) antibodies (Hemagglutination inhibition, HAI) for each treatment arm
Increase in HAI titer against A/California/07/2009 | Day 0 and 30
  Geometric mean fold increase (GMFI) of anti-A/California/07/2009 (H1N1) HAI serum antibodies for each treatment arm
HAI sero-response | Day 0 and 30
  The proportion of participants, regardless of sero-status, within each treatment arm who experience an H1N1 CA/07/2009 specific sero-response post-dose. Sero-response is defined as a ≥4-fold rise in HAI titer from baseline.
Serum IgG response | Day 0 and 30
  The proportion of participants within each treatment arm with a greater or equal to 2-fold rise in serum lgG antibody responses to whole virus CA/07/2009 by ELISA
Increase in serum IgG | Day 0 and 30
  Geometric mean fold increase (GMFI) within each treatment arm in serum lgG antibody responses to whole virus CA/07/2009 by ELISA
Serum IgA response | Day 0 and 30
  The proportion of participants within each treatment arm with a greater or equal to 2-fold rise in serum lgA antibody responses to whole virus CA/07/2009 by ELISA
Increase in serum IgA | Day 0 and 30
  Geometric mean fold increase (GMFI) within each treatment arm in serum lgA antibody responses to whole virus CA/07/2009 by ELISA
Salivary IgA Response | Day 0 and 30
  The proportion of participants within each treatment arm with a greater or equal to 2-fold rise in salivary lgA antibody responses to whole virus CA/07/2009 by ELISA
Increase in salivary IgA | Day 0 and 30
  Geometric mean fold increase (GMFI) within each treatment arm in salivary lgA antibody responses to whole virus CA/07/2009 by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Q-Pharm Pty Limited, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No